CLINICAL TRIAL: NCT00230828
Title: Patient-reported Outcomes With Bifeprunox or Olanzapine in the Treatment of Schizophrenia. A Pharmacoeconomic Study Carried Out in Connection With the S1543003 And S1543004 Clinical Trials
Brief Title: Patient-reported Outcomes in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S154.3.005
Record Dates: First submitted 2005-09-12; First posted 2005-10-03 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox

INTERVENTIONS:
Drug: bifeprunox

SUMMARY:
Patient-reported health economic outcomes for patients enrolled in S1543003 and S1543004 protocols

ELIGIBILITY:
Inclusion Criteria:

* Participate in S1543003 and S1543004 in the U.S. sites

Exclusion Criteria:

* Participate in S1543003 and S1543004 other than U.S. sites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05; Primary Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals